CLINICAL TRIAL: NCT03854448
Title: The Incidence and Predictors of Developing Atrial Fibrillation in Patients With Inferior ST-segment Elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, ahmed atef ahmed atef, principal investigator, Assiut University
Other Study IDs: AF in inferior STEMI after PCI
Record Dates: First submitted 2019-02-24; First posted 2019-02-26 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation
Keywords: inferior STEMI
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography, Ambulatory; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: holter monitoring — Transthoracic Echocardiography (TTE) Left atrial ( LA) volume will be measured using standard apical two- and four-chamber views on the frame just prior to mitral valve opening and as specified by current American Society of Echocardiography guidelines (10) LA volume is indexed to body surface area. Mitral inflow velocity is obtained in the apical four-chamber view by placing a pulsed-Doppler sample volume between the tips of the mitral leaflets. Mitral annular velocity is assessed during the early phase of diastole(e=) using pulsed-wave Doppler sampling of septal mitral annular motion from the four chamber view.
  24 to 48 hours Holter monitoring after 1 month after PCI
  Other Names: echocardiography

SUMMARY:
Is to analyze the incidence and predictors of developing AF in patients with inferior infarction who undergo PCI with and without atrial and SN branches occlusion

DETAILED DESCRIPTION:
Atrial fibrillation (AF) occurs in 5% to 18% of patient with acute ST-segment elevation myocardial infarctions (STEMIs) and 4.5% in patients with STEMI treated with percutaneous coronary intervention (PCI).

Diagnosis of AF in acute myocardial infarction (AMI) patients is important because it increases the risk of cardiovascular event and associated with increased in-hospital and long term rates . Atrial ischemia/infarction translates into P Q segment depression or elevation on the electrocardiogram and often associates with atrial tachyarrhythmias .

Side-branch obstruction is one of the adverse effects of PCI the location of the culprit vessel also affects the occurrence of AF in AMI Atrial arteries arise from the right coronary artery (RCA) and circumflex coronary artery (CX) and extend through the atrial myocardium to supply both chambers It is therefore conceivable that PCI of lesions located at the RCA and CX could lead to an accidental atrial branch occlusion .

Atrial myocardial ischemia secondary to atrial branches occlusion (ABO) might lead to mechanical atrial dysfunction, increased electrical vulnerability to atrial arrhythmias, and late structural remodeling .

The sino nodal (SN) artery originates from the proximal portion of the RCA in about 60% of humans Side branch occlusion of the SN artery occurring accidentally during PCI for proximal RCA lesions would provide an opportunity to produces SN dysfunction in humans. Uptill now , there have been no systematic studies concerning SN dysfunction caused by side-branch occlusion of the SN artery during PCI .

Left atrial volume seems to be a strong predictor of incident of AF , with increase in left atrial filling pressures, atrial stretch and enlargement of the chamber occur, leading to remodeling of the structure, physiologic properties, and electrical milieu of the left atrium, culminating in the development of AF

ELIGIBILITY:
Inclusion Criteria:

* Patients with inferior STEMI who will undergo PPCI (primary percutaneous coronary intervention )

Exclusion Criteria:

* -A history of preexisting AF
* Prior documentation of heart failure or reduced left ventricular ejection fraction < 50%,
* Severe valvular disease ( rheumatic , sclerotic ) or secondary to AMI
* Left ventricular hypertrophy : enlargement and thickening of the walls of the ventricle
* Patients with inferior STEMI treated with intravenous thrombolysis or conservative strategy
* Patients with inferior STEMI who undergo primary PCI and associated with right ventricular or posterior infarction
* History of pulmonary embolism or COPD ( chronic obstructive pulmonary disease )
* Those with thyrotoxicosis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with inferior S-T elevation myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
incidence of atrial fibrillation in inferior STEMI patients after primary Percutaneous Coronary Intervention | baseline
  incidence of atrial fibrillation in inferior STEMI patients after primary Percutaneous Coronary Intervention

SECONDARY OUTCOMES:
atrial branches occlusion and left atrial volume index as predictors of atrial fibrillation | baseline
  atrial branches occlusion and left atrial volume index as predictors of atrial fibrillation in inferior STEMI patients after primary Percutaneous Coronary Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Yehia Taha Kishk kishk, MD, Study Chair — Professor of cardiology department Assiut University; Mohamed Ali Mohamed Tohamy tohamy, MD, Study Director — Lecturer of cardiology department Assiut University

REFERENCES:
- See also: Clinical factors associated with the development of atrial fibrillation in the year following STEMI treated by primary PCI — https://www.ncbi.nlm.nih.gov/pubmed/?term=Clinical+factors+associated+with+the+development+of+atrial+fibrillation+in+the+year+following+STEMI+treated+by+primary+PCI
- See also: Impact of atrial fibrillation in patients with ST-elevation myocardial infarction treated with percutaneous coronary intervention — https://www.ncbi.nlm.nih.gov/pubmed/24176066
- See also: Acute regional left atrial ischemia causes acceleration of atrial drivers during atrial fibrillation — https://www.ncbi.nlm.nih.gov/pubmed/23454487
- See also: Atrial coronary artery occlusion during elective percutaneous coronary angioplasty — https://www.ncbi.nlm.nih.gov/pubmed/23994037
- See also: Sinus arrest caused by occlusion of the sinus node artery during percutaneous coronary intervention for lesions of the proximal right coronary artery — https://www.ncbi.nlm.nih.gov/pubmed/?term=Sinus+arrest+caused+by+occlusion+of+the+sinus+node+artery+during+percutaneous+coronary+intervention+for+lesions+of+the%0Bproximal+right+coronary+artery
- See also: Left Atrial Volume: Important Risk Marker of Incident Atrial Fibrillation — https://www.ncbi.nlm.nih.gov/pubmed/?term=Left+Atrial+Volume%3A+Important+Risk+Marker+of+Incident+Atrial+Fibrillation
- See also: Coronary artery disease affecting the atrial branches is an independent determinant of atrial fibrillation after myocardial infarction — https://www.ncbi.nlm.nih.gov/pubmed/?term=Coronary+artery+disease+affecting+the+atrial+branches+is+an%0Bindependent+determinant+of+atrial+fibrillation+after+myocardial+infarction
- See also: Electrophysiological Effects of Selective Atrial Coronary Artery Occlusion in Humans — https://www.ncbi.nlm.nih.gov/pubmed/27151531
- See also: Long Term Prognosis of Atrial Fibrillation in ST-Elevation Myocardial Infarction Patients Undergoing Percutaneous Coronary Intervention — https://www.ncbi.nlm.nih.gov/pubmed/28390742
- See also: Left Atrial Size : Physiologic Determinants and Clinical Applications — https://www.ncbi.nlm.nih.gov/pubmed/?term=Left+Atrial+Size%0BPhysiologic+Determinants+and+Clinical+Applications